CLINICAL TRIAL: NCT04953832
Title: Neurotherapeutics as an Adjunctive Approach to Enhance Exposure Outcomes in Anxiety
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Jessica Bomyea, Assistant Professor, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 191018
Record Dates: First submitted 2021-06-21; First posted 2021-07-08 (Actual); Last update posted 2021-10-01 (Actual); Status verified 2021-09

CONDITIONS: Anxiety Disorders
MeSH Terms: conditions — Anxiety Disorders | interventions — Cognitive Training

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cognitive Training + exposure (Experimental): Participants will complete adaptive computerized cognitive training plus a series of speech tasks
  Interventions: Behavioral: Cognitive Training
- No training + exposure (Active Comparator): Participants will complete a low-dose computerized cognitive program plus a series of speech tasks
  Interventions: Behavioral: Cognitive Training

INTERVENTIONS:
Behavioral: Cognitive Training — Participants are asked to remember a series of items while solving puzzles.

SUMMARY:
Anxiety disorders are highly prevalent and costly to the individual and society. Exposure-based cognitive behavioral therapy (CBT) is the gold-standard intervention for anxiety disorders, although this approach does not fully reduce symptoms for all individuals. Therefore there is a need for innovative intervention approaches. One approach to augment and improve existing therapies would be to enhance the neurocognitive basis of fear extinction processes, which are the model on which treatments are based. Enhancing these processes may be possible through computerized cognitive training techniques which target executive functioning, the cognitive processes that help people manage complex cognitive activities. The proposed project is a proof-of-concept pilot study investigating the potential for training of executive functioning to improve anxiety-related outcomes. Individuals with elevated levels of social anxiety will be randomized to single-session COGnitive Enhancement Training (COGENT) or sham training program (ST). All participants will complete a single speech session where they present three 7-minute impromptu speeches and rate their anxiety at specific intervals. Participants will then complete the COGENT paradigm and affective processing task while undergoing fMRI.

ELIGIBILITY:
Inclusion Criteria:

1. Screened positive for anxiety symptoms
2. Between the ages of 18-55, inclusive.
3. Have signed informed consent document(s) indicating that he/she understands the purpose of and procedures required for the study and is willing to participate in the study.
4. Have sufficient proficiency in English language to understand and complete interviews, questionnaires, and all other study procedures.

Exclusion Criteria:

1. Evidence of psychosis, bipolar disorder, or severe substance use disorder based on clinical cutoffs on self report measures
2. Current neurological conditions based on brief medical history
3. Current psychotherapy for anxiety or psychotropic medications
4. MRI contraindications including: cardiac pacemaker, metal fragments in eyes/skin/body (shrapnel), aortic/aneurysm clips, prosthesis, by-pass surgery/coronary artery clips, hearing aid, heart valve replacement, shunt (ventricular or spinal), electrodes, metal plates/pins/screws/wires, or neuro/bio-stimulators (TENS unit), persons who have ever been a metal worker/welder, history of eye surgery/eyes washed out because of metal, vision problems uncorrectable with lenses, inability to lie still on one's back for 60 minutes; prior neurosurgery; tattoos with metal dyes, unwillingness to remove body piercings, and pregnancy.
5. Active suicidal ideation endorsed on the depression self-report measure.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2021-09-01 (Actual); Study Completion 2021-09-01 (Actual)

PRIMARY OUTCOMES:
BOLD activation during cognitive task | immediately after the intervention
  Working Memory Span task during fMRI
BOLD activation during emotional task | immediately after the intervention
  Face processing task during fMRI

SECONDARY OUTCOMES:
Speech anxiety ratings | baseline, ratings during 3 speeches
  Subjective units of distress, scaled from 0 to 100, during each of 3, 7-minute speech activities

CONTACTS AND LOCATIONS:
Locations (1):
- UC San Diego, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No